CLINICAL TRIAL: NCT02525991
Title: A Phase IV, Open-label, Non-randomized, Clinical Trial to Evaluate the Safety of Self-administered ADASUVE® (Staccato Loxapine for Inhalation) in Agitated Patients Outside the Hospital Setting
Brief Title: Phase IV to Evaluate the Safety of Self-administered ADASUVE® in Agitated Patients Outside the Hospital Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-Loxapine-2015-01
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Agitation
Keywords: schizophrenia; bipolar disorder
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Intervention: treatment with Loxapine staccato- just one treatment arm - outside the hospital setting.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staccato® Delivery System Loxapine (Experimental): Staccato® Delivery System Loxapine, 9.1 mg one dose
  Interventions: Device: Staccato® Delivery System Loxapine (ADASUVE®)

INTERVENTIONS:
Device: Staccato® Delivery System Loxapine (ADASUVE®) — one dose Loxapine Staccato 9.1 mg
  Other Names: ADASUVE®

SUMMARY:
Phase IV, multinational, multicentre, open-label, non-randomized, clinical trial conducted in Europe (Spain, Germany, Finland, Norway, Romania and Austria) to evaluate the safety profile of ADASUVE® in agitated patients with schizophrenia or bipolar disorder when self-administered outside of a hospital setting without the supervision of a healthcare professional. The Study will aim to include approximately 500 patients who have been previously treated with ADASUVE® in the last 6 months prior to screening or recently treated during the planned recruitment period of 6 months with a 'positive outcome' ('ADASUVE® responder') according to Clinical Global Impressions (CGI-I) scale, from a total of about 30-34 centers. All patients will be followed up for a maximum of 6 months from baseline, during which it is expected that a new episode of agitation will occur.

DETAILED DESCRIPTION:
OVERALL STUDY DESIGN:

This is a phase IV, multinational, multicentre, open-label, non-randomized, clinical trial conducted in Europe (Spain, Germany, Finland, Norway, Romania and Austria) to evaluate the safety profile of ADASUVE® in agitated patients with schizophrenia or bipolar disorder when self-administered outside of a hospital setting without the supervision of a healthcare professional.

The Study will aim to include approximately 500 patients who have been previously treated with ADASUVE® in the last 6 months prior to screening or recently treated during the planned recruitment period of 6 months with a 'positive outcome' ('ADASUVE® responder') according to Clinical Global Impressions (CGI-I) scale, from a total of about 30-34 centers. An 'ADASUVE® responder' is defined as having a CGI-I score at 2 hours after administration of either a 1 (very much improved) or 2 (much improved). All patients will be followed up for a maximum of 6 months from baseline, during which it is expected that a new episode of agitation will occur.

Centers will be selected and qualified primarily based on their estimated number of eligible patients. The patients attending a hospital setting, such as Hospital Wards, Emergency Rooms, Day Care Units, Hospital Home-care units, or other Institutions for an agitation episode treatment will be recruited.

Site study staff will screen patients for potential participation on the clinical study at the time of presentation in a hospital setting for an on-going agitation episode during the recruitment period of 6 months, or retrospectively for a previous one episode within the 6 months prior to screening. The study staff will review the patient's medical records in detail to determine eligibility.

There will be a baseline hospital visit within 2 to 4 weeks after the screening for all pre-selected patients. This hospital visit will be scheduled after the resolution of the episode in patients pre-selected during an on-going agitation episode. Patients with a previous agitation episode will be called by phone by site staff for ensuring that they meet the eligibility requirements for enrolling and planning a baseline visit.

At screening patients and family (or caregivers) will be informed by the study staff that at the baseline visit they will receive a specific training session for the proper self-administration of ADASUVE® outside the hospital setting and about other procedures related to the study.

At the baseline visit, selected patients will be asked to provide the signed informed consent for inclusion in the study before any study related procedures.

Once the informed consent has been obtained the eligibility criteria will be confirmed (including a negative result of the urine pregnancy test performed in women of childbearing potential and that the family member or other caregiver support is in place) for the patient inclusion.

Once the patient is included in the study:

* He/she will receive one unit of ADASUVE® for treating the next agitation episode outside the hospital setting (plus a short-acting beta-agonist bronchodilator for treatment of possible severe respiratory side effects [i.e bronchospasm]).
* Patients with the presence of a family member or other caregiver will receive a specific training session for properly self-administration of ADASUVE® outside the hospital setting and clear indications to identify the appearance of an agitation crisis, based on the recognition of their escalating symptoms experienced in previous agitation episodes.
* Additional educational material will be provided to the patients in a document including:

  o Patient information card for recognition of symptoms of agitation, instructions of the study, information for recognition of respiratory symptoms and instruction of use of the medicine to treat them.
* The patient's diary card will be also delivered to the patient (and family member/caregiver).
* Patient will be trained to use the patient' diary card to register the agitation episode information.

Each patient included in the study will receive a study kit containing: one unit ADASUVE® for the next agitation episode (plus a short-acting beta-agonist bronchodilator as rescue medication to treat severe respiratory symptoms), the instructions for the use of ADASUVE®, ADASUVE® storage instructions, the patient's diary card and the educational material. The patient's kit will also include useful instructions of ADASUVE® storage such as to store locked in a cool, dry place away from direct sunlight, to keep it out of reach of children, not to use it after the expiry date which is stated on the product label, not to discard it in the household waste and to keep it in pouch until time of use.

At baseline the following data will be obtained retrospectively from medical records for each patient and will be recorded in the electronic case report forms: demographics, diagnosis, agitation information of current/previous episode (date/time of the onset, time to improvement and patient status rate at 2h of ADASUVE® administration [CGI-I scale]), respiratory disease history and risks factors, co morbidities/medical history (non-respiratory), concomitant medications, previous ADASUVE® treatment (date and dosing data).

During the 6-month follow-up from baseline visit study staff will conduct a 10-minutes phone-calls (every 3 months approximately) to the enrolled patients or their family member/caregiver. Patients (or family member/caregiver) will be asked for general patient health status. In addition, patients will be reminded to return the medication if they have not presented a new episode of agitation after the 6 months of follow-up from the baseline visit. All these patients will be scheduled for the study staff for an end of study visit with the aim to return the unused study kit. These patients will be excluded from the study. All this related information will be recorded in the electronic case report forms.

Three clinical scenarios can occur following the self-administration of ADASUVE® outside the hospital setting for the treatment of an acute agitation episode:

• If there is an improvement within 2-hours post-dose self-administration of ADASUVE® outside the hospital setting and once the episode of acute agitation has dismissed, the following data will be collected at patient's diary card with adequate family (or caregiver) support:

o Date of the diary completion, person who completed the diary (patient, relatives or caregiver), date/time of the onset of current episode of agitation, date/time of ADASUVE® self-administration, , severity of the episode (CGI-S scale) before ADASUVE® administration and time/rate to improvement of current episode of agitation (CGI-I scale) scores at 2, 10, 20, 30, 60 and 120 minutes after ADASUVE® administration, AEs related to ADASUVE® during the following 24 hours of the self-administration, medications to treat ADASUVE® treatment-emergent AEs (e.g., short-acting bronchodilator) and another medication used following 24 hours of ADASUVE® administration.

Once ADASUVE® treatment has taken place, immediately patient (or a family member/caregiver) must inform the corresponding study investigator to schedule a follow-up hospital visit (within 24-72h after ADASUVE® self-administration). The 24-72h follow-up visit after ADASUVE® self-administration with the study investigator will include a review of data from patient diary card that will be recorded in the electronic case report forms by the investigator staff. Additionally, the study investigator will confirm during the visit that the patient is in good general health based on their judgment and patients will be asked to evaluate their treatment satisfaction after self-administered ADASUVE® outside the hospital setting using a 5-point Likert scale.

* If there is no improvement or worsening of the agitation after 1 hour of ADASUVE® self-administration outside the hospital setting, the patient must attend the assigned hospital for a 2nd dose of ADASUVE® (≥ 2 hours after dose one) or another medication to treat the agitation episode, at the discretion of the investigator. If additionally, the patient had reported an AE after the first administration of ADASUVE® outside the hospital setting and a second dose of ADASUVE® cannot be administered, another medication should be dispensed at hospital setting to treat this agitation episode.
* If after ≥2 hours of ADASUVE® self-administration outside the hospital setting there is a worsening of the agitation episode (once there was a previous improvement within 2-hours post-dose administration), the patient must attend the assigned hospital for a 2nd dose of ADASUVE® or another medication to treat the agitation episode, at the discretion of the investigator.

The following data until discharge will be collected in the electronic case report forms by study staff if there is no improvement or worsening after self-administration of ADASUVE® for patients attending the hospital:

* Other treatments administered for agitation episode in addition to 1st dose of ADASUVE® self-administered outside the hospital setting or to the 2nd dose of ADASUVE® at hospital administration for non-responders patients (number and timing of doses administered)
* Other treatments administered for agitation in addition to 2nd dose of ADASUVE®.
* Date/time of the onset of current episode of agitation
* Time to onset of improvement of current episode
* AEs related to ADASUVE®
* Medications and/or interventions to treat ADASUVE® treatment-emergent AEs
* Status at discharge (admission to hospital, discharge to home or other facility, ongoing hospitalization, leave against medical advice, other) All these patients who self-administered ADASUVE® outside the hospital setting should return the used study kit at the scheduled visit accordingly.

Furthermore, patients will receive a follow-up call at 30 days after the self-administration of ADASUVE® outside the hospital setting to record the general health status of the patient including information about any other AEs related to ADASUVE® experienced during this period.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18-65 years, inclusive
2. Patients (or legal representative) willing and able to provide written Informed Consent Form.
3. Psychiatric patients already diagnosed of schizophrenia or bipolar disorder, according to the Diagnostic and Statistical Manual of Mental Disorders- IV, Diagnostic and Statistical Manual of Mental Disorders- V or International Code of Disease criteria.
4. Patients with an on-going agitation episode, or with a previous one within the 6 months prior to screening, attended and managed in the hospital setting.
5. Previously treated with ADASUVE® with a positive outcome (responders) according to (CGI-I) scale (defined as having a CGI-I score of 1 or 2 at 2 hours after administration of the inhalation)
6. Patients free of active respiratory disease such as acute respiratory signs/symptoms (e.g., wheezing) or with active airways disease (asthma, chronic obstructive pulmonary disease or emphysema).
7. Requirement of family or other caregiver support at study investigator criteria (defined as a patient's relative or caregiver (male or female) ≤ 80 year old, who spend ≥ 3 consecutive hours with patient, with good physical and psychological health status and without physical limitations, reading and writing educational level and able to understand and follow the study procedures).
8. Availability of patient's medical records data about the previous treatment with ADASUVE® at hospital setting.
9. If a female is of childbearing potential and sexually active (except if female is surgically sterile or post-menopausal with history of no menses for at least 24 months), patient must be non-lactating and non-pregnant (with a negative pregnancy test result at baseline visit) and have to agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study.

Exclusion Criteria:

1. Patient diagnosed with dementia.
2. Patients with serious and unstable illnesses including current hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease and congestive heart failure), endocrinologic, neurologic (including stroke, transient ischemic attack, subarachnoidal bleeding, brain tumor, encephalopathy, and meningitis).
3. Patients with a history of allergic reactions to loxapine or amoxapine
4. Patients who have received an investigational drug within 30 days prior to the current agitation episode must be excluded.
5. Patients who are considered by the investigator, for any reason, to be unable to self-administer the inhalation device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Serious adverse events and adverse events of special interest ( respiratory) | one year
  To assess the safety profile of self-administered ADASUVE® outside the hospital setting in a population of patients that are known ADASUVE® responders and well trained on the use of the product, with a primary focus on serious adverse events (SAEs) and adverse events of special interest (AESI) related to ADASUVE®, including respiratory events

SECONDARY OUTCOMES:
time to improvement of the agitation episode after the self-administration of ADASUVE® outside the hospital setting. | one year
  To evaluate the time to improvement of the agitation episode after the self-adminsitration of ADASUVE® outside the hospital setting.
Prevalence of the medication for treating agitation episode in the hospital setting after self-administration of ADASUVE®. | one year
  To determine the prevalence of the medication treatment for an agitation episode in the hospital setting after self-administration of ADASUVE®.

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Teixeira, PharmD, PhD, Study Director — Ferrer Internacional SA
Locations (1):
- Ferrer Internacional S.A., Barcelona, Spain

REFERENCES:
- [Derived] Gil E, Garcia-Alonso F, Boldeanu A, Baleeiro Teixeira T; Loxapine Inhaled Home Use study investigator's team. Safety and efficacy of self-administered inhaled loxapine (ADASUVE) in agitated patients outside the hospital setting: protocol for a phase IV, single-arm, open-label trial. BMJ Open. 2018 Oct 2;8(10):e020242. doi: 10.1136/bmjopen-2017-020242. PMID 30282677